CLINICAL TRIAL: NCT05373563
Title: Quality of Postpartum Cesarean Recovery Score Validity Reliability
Acronym: ObsQoR-11
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, ümmühan kılıç, Principal Investigator, Ondokuz Mayıs University
Other Study IDs: SAMSUN HEALTH DİRECTORATE
Record Dates: First submitted 2022-04-22; First posted 2022-05-13 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Failed VBAC (Vaginal Birth After Cesarean)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cesarean section women — The test will be applied to women who have had a cesarean section and the Turkish validity and reliability of the scale will be determined according to the answers given.

SUMMARY:
In order to provide the best care of patients after cesarean section, to help solve all their biopsychosocial problems in the recovery process, and to shorten the hospitalization period, it should be measured with appropriate measurement tools for various evaluations. The Scale of Post-cesarean Healing Quality You will provide in adapting the ObsQoR-11 questionnaire to Turkish.

DETAILED DESCRIPTION:
In order to provide the best care of patients after cesarean section, to help solve all their biopsychosocial problems in the recovery process, and to shorten the hospitalization period, it should be measured with appropriate measurement tools for various evaluations. We will provide the Scale of Post-Cesarean Healing Quality in adapting the ObsQoR-11 questionnaire to Turkish.It is important to define well the recovery after cesarean section.

ELIGIBILITY:
Inclusion Criteria:

* Must be Over 18 age,
* Must be literate women,
* Must be no neurological disease

Exclusion Criteria:

* Must be unwilling to participate in the study
* Must be under 18 years old women

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Study study of 18 patients using large cesarean section.
Study Population: Study study of 18 patients using large cesarean section.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2022-07-24 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Quality of Postpartum Cesarean Recovery Score validity reliability | July 2022-October 2022
  Measuring early recovery after cesarean section
obstetric qualityof- recovery score (ObsQoR-11) | About six mount
  Women were approached while in the postnatal ward 24 h after CS and asked to complete the ObsQoR-11K questionnaire and to choose a point in the 100-mm numeric rating scale (NRS) to evaluate global health status. Women rated each recovery item using an 11-point numerical Likert scale (0 = strongly negative; 10 = strongly positive).
  Global health status was measured using NRS indicated by a 100 mm line (0 = 'worst imaginable health status' and 'sad' face; 100 = 'best imaginable health status' and 'happy' face).

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Kıymaz,, PhD, Principal Investigator — Samsun Provincial Health Directorate; Esra Saraçoğlu, PhD, Study Chair — Samsun Provincial Health Directorate
Locations (1):
- Samsun Health Directorate, Samsun, Black Sea, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No